CLINICAL TRIAL: NCT04528498
Title: The Embryo Health Study: Prospective Longitudinal Analysis of PGT-P
Brief Title: Embryo Health Study
Acronym: EHS
Status: Recruiting | Type: Observational
Sponsor: Genomic Prediction Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Genomic Prediction Inc 616
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2024-08

CONDITIONS: Infertility; Hereditary Diseases
MeSH Terms: conditions — Infertility; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Amplified DNA from trophectoderm biopsies of human embryos and from saliva samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Preimplantation Genetic Testing — Embryo biopsies will undergo preimplantation genetic testing for aneuploidies as per standard of care, and polygenic disease risk (PGT-P) will be computed for these samples.

SUMMARY:
This study intends to determine the patients' perception and motivation to obtain additional information on their preimplantation embryos' risks of polygenic disorders. Patients undergoing IVF and genetic testing on their embryos for aneuploidies will be given the option to obtain information of their embryos' polygenic disease risk after receiving genetic counseling.

DETAILED DESCRIPTION:
Patients planning to use PGT-A and who meet the inclusion criteria will be offered participation by their IVF physician prior to initiating cycle stimulation. Eligible and interested patients will be contacted, counseled and consented for participation in the study by a Genetic Counselor at Genomic Prediction Clinical Laboratory. This will include genetic counseling to address the benefits and limitations of PGT-A and PGT-P, the family history of diseases currently tested under PGT-P, what diseases they may be interested in testing, the process of obtaining saliva samples, and the information provided by PGT-P results.

A total of 500 patients will complete the study and may be recruited from any IVF clinic in the United States. After being enrolled in the study, patients will have two options. One option is to receive PGT-A results first and then decide if they wish to receive the PGT-P results. A second option is to receive a single comprehensive report. All patients will receive a report indicating the predicted karyotype of each embryo (PGT-A) and, according to which option they elected, may also receive a report on any or all of the following elected diseases: Type 1 Diabetes, Type 2 Diabetes, Coronary Artery Disease, Heart Attack, Hypercholesterolemia, Hypertension, Testicular Cancer, Prostate Cancer, Malignant Melanoma, Breast Cancer, Basal Cell Carcinoma. Furthermore, a genetic ancestry test will be performed on each submitted saliva sample to determine potential PGT-P performance and which disease predictors can be computed based on the patients ethnic background.

ELIGIBILITY:
Inclusion Criteria:

* All couples of Caucasian or East Asian ancestry above the age of 18 who elect to have PGT-A as part of their IVF treatment cycle.

Exclusion Criteria:

* Any case where biological parental DNA is unavailable.
* Any case involving PGT-M or PGT-SR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing IVF with preimplantation genetic testing for aneuploidies (PGT-A).
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Patients' interest in Preimplantation Genetic Testing for Polygenic Disorders | 2 years
  Patients' interest in obtaining information on their embryos' polygenic disease risk will be measured in a scale of 1-5. 1 being "Not interested" and 5 "highly interested".

CONTACTS AND LOCATIONS:
Locations (1):
- Genomic Prediction Clinical Laboratory, North Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data will be available after publication of the study main findings, either as supplemental material or in a public data repository.